CLINICAL TRIAL: NCT04286321
Title: Achieving Nutritional Adequacy Of Vitamin K With An Egg/Plant-Based Food Pairing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Richard Bruno, Professor and Principal Investigator, Ohio State University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2019H0504-B
Record Dates: First submitted 2020-02-22; First posted 2020-02-27 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Nutritional Requirements
Keywords: Vitamin K; Egg; Spinach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Zero hard-boiled egg (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested alone prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Zero hard-boiled egg at 0 h
- One hard-boiled egg at 0 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested along with one hard-boiled egg prior to the 72-h pharmacokinetics trial.
  Interventions: Other: One hard-boiled egg at 0 h
- Two hard-boiled eggs at 0 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested with two whole eggs (9.6 g fat) prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Two hard-boiled eggs at 0 h
- Three hard-boiled eggs at 0 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested along with three hard-boiled eggs prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Three hard-boiled eggs at 0 h
- One hard-boiled egg at 3 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested alone at 0 h prior to the 72-h pharmacokinetics trial followed by one hard-boiled egg 3 hours after spinach consumption.
  Interventions: Other: One hard-boiled egg at 3 h
- One hard-boiled egg at 0 h + One hard-boiled egg at 3 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested along with one hard-boiled egg at 0 h prior to the 72-h pharmacokinetics trial followed by one egg 3 hours after spinach consumption.
  Interventions: Other: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
- Two egg whites at 0 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested along with two egg whites prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Two egg whites at 0 h
- Vegetable oil at 0 h (Experimental): Deuterium-labeled spinach containing 500 μg PQ will be ingested along with 9.6 grams of vegetable oil prior to the 72-h pharmacokinetics trial.
  Interventions: Other: Vegetable oil at 0 h

INTERVENTIONS:
Other: Zero hard-boiled egg at 0 h — No eggs will be consumed on test day along with spinach consumption
  Arms: Zero hard-boiled egg
Other: One hard-boiled egg at 0 h — One egg will be consumed on test day along with spinach consumption
  Arms: One hard-boiled egg at 0 h
Other: Two hard-boiled eggs at 0 h — Two eggs will be consumed on test day along with spinach consumption
  Arms: Two hard-boiled eggs at 0 h
Other: Three hard-boiled eggs at 0 h — Three eggs will be consumed on test day along with spinach consumption
  Arms: Three hard-boiled eggs at 0 h
Other: One hard-boiled egg at 3 h — One egg will be consumed on test day three hours after spinach consumption
  Arms: One hard-boiled egg at 3 h
Other: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h — Two eggs will be consumed on test day: one along with spinach consumption and the other one three hours after spinach consumption
  Arms: One hard-boiled egg at 0 h + One hard-boiled egg at 3 h
Other: Two egg whites at 0 h — Two egg whites will be consumed on test day along with spinach consumption
  Arms: Two egg whites at 0 h
Other: Vegetable oil at 0 h — 9.6 grams of Vegetable oil will be consumed on test day along with spinach consumption
  Arms: Vegetable oil at 0 h

SUMMARY:
Malnutrition of the fat-soluble nutrient vitamin K (phylloquinone; PQ) is problematic. Since PQ is rich in plant foods (e.g. spinach) that are mostly absent of accessible lipid, dietary patterns that can potentiate PQ bioavailability by pairing vegetables with lipid-rich foods have been emphasized. The purpose of this study is to use deuterium-labeled spinach (containing stable isotopes of PQ) to validate eggs as a dietary tool to improve PQ bioavailability directly from a model plant food, and hence achieve nutrient adequacy. It is expected that compared with deuterium-labeled spinach alone, co-ingestion of eggs will increase plasma bioavailability of spinach-derived deuterium-labeled PQ without affecting time to maximal concentrations or half-lives. Further, phospholipid-rich egg yolk lipid will enhance nutrient bioavailability compared with vegetable oil. The outcomes will serve as the foundation for easy-to-implement message of public health importance in support of whole eggs and egg whites as part of a plant-based dietary pattern.

DETAILED DESCRIPTION:
In the US, 43-63% of men and women do not meet recommended intakes for PQ. Dietary recommendations strongly encourage a diet rich in fruits and vegetables to meet dietary PQ requirements. However, PQ bioavailability from most plant foods is quite poor, thereby emphasizing a need for effective food pairings that can enhance the absorption and promote adequate status of these health-promoting nutrients. The objective of this study is to demonstrate that an effective food pairing of spinach with phospholipid lipid-rich eggs promotes intestinal absorption of spinach-derived PQ, and hence achieve nutrient adequacy. Our hypothesis is that the bioavailability of PQ from deuterium-labeled spinach will be potentiated by egg intake in a dose-dependent manner by increasing their secretion in intestinal-derived chylomicrons. Furthermore, phospholipid-rich whole eggs will enhance spinach-derived PQ bioavailability compared with vegetable oil, and will be most functionally responsible for the benefits of eggs to enhance nutrient absorption. Additionally, egg whites will more greatly promote nutrient bioaccessibility compared with spinach alone.

To test this, our specific aim is to assess egg-mediated improvements in PQ bioavailability by conducting a cross-over pharmacokinetic study in healthy men and women. In Study Arms 1-4, participants will ingest deuterium-labeled spinach (containing 500 μg PQ) with 0, 1, 2, or 3 hardboiled eggs (containing 0, 4.8, 9.6, or 14.4 g total fat, respectively). In Study Arm 5, participants will ingest spinach alone followed by 1 egg 3-hours later. In Study Arm 6, participants will ingest spinach with 1 egg followed by another egg 3-hours later. In Study Arm 7, participants will ingest spinach with two egg whites. In Study Arm 8, participants will ingest spinach with 9.6 grams of vegetable oil. Thus, Study Arms 1-4 will test the dose-dependent effects of eggs on PQ bioavailability, Study Arms 5-6 (with comparison to Study Arms 1 and 2) will test the 'timing'-dependent effects of eggs on PQ bioavailability, and Study Arms 7-8 will test the matrix effect on PQ bioavailability. Eucaloric diets will be controlled for PQ intakes for 3 d prior to and during the initial 24 h of each trial to minimize heterogeneity of pharmacokinetic responses. Spinach-derived deuterium-labeled PQ will be measured in plasma and isolated chylomicrons collected at timed intervals from 0-72 h post-meal ingestion, and biomarkers of antioxidant status and oxidative distress will be assessed at baseline (0 h) of each trial. Outcomes from this study are expected to establish that egg lipids substantially enhance plant-derived PQ bioavailability (based on AUC0-72 h, Cmax, and % estimated absorption) independent of any changes in oxidative distress.

The rationale for this study is that, by establishing the efficacy of eggs and egg yolk lipids to potentiate plant-derived fat-soluble nutrient bioavailability, a strong framework will exist for an easily implementable health-promoting food pairing strategy to overcome malnutrition of PQ.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) = 19-25 kg/m2
* Normolipidemic (total cholesterol <240 mg/dL; triglyceride <150 mg/dL)
* Fasting glucose <100 mg/dL
* Normal hematocrit level (41%-50% for men and 36%-48% for women)
* Normal hemoglobin level (13.5-17.5 g/dL for men and 12.0-15.5 g/dL for women)
* No use of dietary supplements for >1 month
* No use of medications that affect lipid or glucose metabolism
* Non-smoker
* No history of gastrointestinal disorders

Exclusion Criteria:

* Egg allergy
* Alcohol intake > 2 drinks per day
* Aerobic activity >7 h/wk
* Body mass change >2 kg in the past 1 month
* Women who are pregnant, lactating, or initiated or changed birth control in the past 3 month
* Vegetarian

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Vitamin K Bioavailability | 0, 3, 4.5, 6, 7.5, 9, 12, 24, 36, 48, 72 hours post-ingestion of spinach
  Area under the curve of deuterium-labeled phylloquinone

SECONDARY OUTCOMES:
Vitamin K Tmax | 0-72 hours post-ingestion of spinach
  Time to reach maximum plasma concentration of deuterium-labeled phylloquinone
Chylomicron Vitamin K | 0, 3, 4.5, 6, 7.5, 9, 12 hours post-ingestion of spinach
  Deuterium-labeled phylloquinone concentration in chylomicron
Estimated Absorption (%Dose) of Vitamin K | 0-72 hours post-ingestion of spinach
  Absorption of deuterium-labeled phylloquinone
Vitamin K Cmax | 0-72 hours post-ingestion of spinach
  Maximum plasma concentration of deuterium-labeled phylloquinone
Elimination Rate of Vitamin K | 0-72 hours post-ingestion of spinach
  Rate of plasma elimination of deuterium-labeled phylloquinone

CONTACTS AND LOCATIONS:
Overall Officials: Richard Bruno, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- Bruno Lab, Columbus, Ohio, United States